CLINICAL TRIAL: NCT04318431
Title: Prevalence of SARS -Cov2 Carriage in Asymptomatic and Mildly-symptomatic Children, a Cross-sectional, Prospective, Multicentre, Observational Study in Primary Care.
Brief Title: Prevalence of SARS -Cov2 Carriage in Asymptomatic and Mildly-symptomatic Children
Acronym: COVILLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: Association Clinique Thérapeutique Infantile du val de Marne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: COVILLE; 2020-A00724-35 (Other: ID-RCB)
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Covid19
Keywords: Sars-Cov2 rhino-pharyngeal carriage; primary care; children
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Data collection and rhinopharyngeal swab (Other): After information, the collection of consent will be carried out. A clinical information sheet will be completed by the investigator in order to collect socio-demographic data, history, clinical symptoms and signs, and complementary examinations performed.
  During the same consultation, a rhinopharyngeal swab will be taken for the detection of SARS -Cov2 and other respiratory pathogens by PCR.
  Interventions: Diagnostic Test: Data collection and rhinopharyngeal swab

INTERVENTIONS:
Diagnostic Test: Data collection and rhinopharyngeal swab — Testing for SARS -Cov2 and other respiratory pathogens by PCR via nasopharyngeal swabbing and IgM/IgG rapid serology
  Other Names: IgM/IgG rapid serology

SUMMARY:
This study is expected to provide, for the first time, data on Cov2-SARS circulation in asymptomatic children and children with moderate respiratory symptoms in order to construct the severity pyramid of this novel pathogen. This information will be essential in the coming weeks to understand the dynamics of the transmission of this pathogen at the population level and to highlight the relevance of public health interventions, particularly with regard to the systematic closure of schools and childcare facilities.

DETAILED DESCRIPTION:
Cov2-SARS is an emerging respiratory virus of the coronavirus family responsible for a global epidemic since November 2019. As of March 10, 2020, it had caused more than 160,000 cases of corona virus disease (COVID-19), including more than 6,500 deaths worldwide. France is one of the main epidemic outbreaks with more than 5,000 confirmed cases and the number of diagnosed patients is increasing every day.

The number of confirmed paediatric cases is relatively low, and the mortality rate in children is close to zero. This contrast suggests that children are more likely to present pauci-symptomatic or even asymptomatic forms of the disease, which are therefore undiagnosed in most cases. Given the rapid spread of this virus, and the fact that indigenous cases without an obvious chain of transmission now appear to be frequent in France, it is possible that the pauci-symptomatic or asymptomatic child may play a role in the transmission of the pathogen and the dynamics of the epidemic, as documented for other respiratory pathogens such as influenza. Based on this hypothesis, the closure of children's communities has been organized in France and other highly endemic countries.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic children:
* Age between birth and 15 years
* Carrying out a visit within the framework defined by the learned societies and professional organisations representative of paediatrics in France, i.e. :
* The consultation of the first month and all consultations involving compulsory vaccinations (2, 4, 5, 11, 12, 16 months).
* Consultations for acute pathologies, infectious or not.
* Monitoring of chronic diseases that warrant clinical examination (the majority of which can be carried out by telemedicine) or in the case of acute exacerbation.
* In one of the participating outpatient centres
* During the study period
* With a clinical examination that does not reveal any progressive infectious pathology

AND Pauci-symptomatic children

* Age between birth and 15 years,
* Consultant at one of the participating outpatient centres
* During the study period
* And presenting with a mild respiratory infection:
* Rhinopharyngitis, Acute otitis media, Angina, Bronchitis, etc.
* Acceptance to participate in the protocol by one of the holders of parental authority
* Affiliated to a social security

Exclusion Criteria:

* Refusal to participate in the study

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 605 (Actual)
Dates: Start 2020-04-14 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Proportion of asymptomatic children or children with mild respiratory symptoms | 14 days
  Proportion of asymptomatic children or children with mild respiratory symptoms (mildly-symptomatic children) with a positive SARS-Cov2 Reverse Transcriptase Polymerase Chain Reaction (RT-PCR) on rhino pharyngeal swab or/and IgM/IgG positive serology in the Ile-de-France region during an epidemic period.

SECONDARY OUTCOMES:
Confirmed Cov2-SARS cases by age | 14 days
  The proportion of confirmed Cov2-SARS cases in mildly-symptomatic and asymptomatic children in different age groups (defined as 6-23 months, 2-4 years, 5-9 years, 10-15 years).
Confirmed Cov2-SARS cases by symptoms | 14 days
  The proportion of confirmed Cov2-SARS cases based on the symptoms presented by the patients
Viral load | 14 days
  The viral load of children with SARS-Cov2 positive Reverse Transcriptase Polymerase Chain Reaction (RT-PCR) depending on the symptoms and the age of the patients
Other respiratory viruses | 14 days
  The proportion of co-infection with other respiratory viruses among children with SARS -Cov2 RT-PCR positive
Sars-Cov2 IgM | 14 days
  Proportion of patients with Sars-Cov2 IgM +
Sars-Cov2 IgG | 14 days
  Proportion of patients with Sars-Cov2 IgG +

CONTACTS AND LOCATIONS:
Locations (22):
- France (22):
  - Cabinet du Dr Belaroussi, Boulogne
  - Cabinet du Dr Derkx, Champigny-sur-Marne
  - Cabinet du Dr Coicadan, Chennevières-sur-Marne
  - 14 Av rené Samuel, Clamart
  - Cabinet du Dr Corrard, Combs-la-Ville
  - 10 rue Delambre, Lagny-sur-Marne
  - 157 Avenue du Général Leclerc, Maisons-Alfort
  - 21 Grande Rue Charles de Gaulle, Nogent-sur-Marne
  - Cabinet du Dr Deberdt, Nogent-sur-Marne
  - Cabinet du Dr Wollner, Nogent-sur-Marne
  - 4 allée des Norottes, Noisy-le-Grand
  - Cabinet du Dr D'acremont, Paris
  - 146 Avenue Ledru Rollin, Paris
  - 132 Boulevard du Montparnasse, Paris
  - Cabinet du Dr Romain, Paris
  - Cabinet du Dr Turberg-Romain, Paris
  - 15 Quai Louis Blériot, Paris
  - Cabinet du Dr Michot, Paris
  - 24 rue Volta, Puteaux
  - Cabinet du Dr Cohen, Saint-Maur-des-Fossés
  - Cabinet de Pédiatrie des Docteurs Ravilly et Bessa, Villejuif
  - 13 Villa Beauséjour, Vincennes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cohen R, Jung C, Ouldali N, Sellam A, Batard C, Cahn-Sellem F, Elbez A, Wollner A, Romain O, Corrard F, Aberrane S, Soismier N, Creidy R, Smati-Lafarge M, Launay O, Bechet S, Varon E, Levy C. Assessment of SARS-CoV-2 infection by Reverse transcription-PCR and serology in the Paris area: a cross-sectional study. BMJ Paediatr Open. 2020 Dec 29;4(1):e000887. doi: 10.1136/bmjpo-2020-000887. eCollection 2020. PMID 33665371